CLINICAL TRIAL: NCT03389204
Title: Upper Limb Function After Breast Cancer Surgery: the Role of Post-operative Physical Therapy Intervention- Randomized Control Trial
Brief Title: Upper Limb Function After Breast Cancer Surgery: the Role of Post-operative Physical Therapy Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assuta Medical Center (Other)
Responsible Party: Principal Investigator, Sergio Gabriel Susmallian, Head of the Department of General Surgery, Assuta Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: AMC2020-17
Record Dates: First submitted 2017-12-26; First posted 2018-01-03 (Actual); Last update posted 2021-01-26 (Actual); Status verified 2021-01

CONDITIONS: Breast Neoplasms
Keywords: Breast surgery; Physiotherapy; Breast Cancer; Shoulder pain; Shoulder motion
MeSH Terms: conditions — Breast Neoplasms; Shoulder Pain | interventions — Physical Therapy Modalities

STUDY DESIGN:
Intervention Model Description: RCT intervention and not intervention
Who Masked: Participant
Masking Description: Participants were blinded to physical support or not
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Breast surgery and exercise (Active Comparator): Patient that underwent breast surgery only without other intervention with exercise of the upper limb and instruction to continue after discharge.
  Interventions: Other: PHYSICAL THERAPY
- Breast surgery and no exercise (Active Comparator): Patient after breast surgery alone are discharged without exercise and instructions.
  Interventions: Other: PHYSICAL THERAPY
- Breast, axilar surgery with exercise (Active Comparator): Patients that underwent surgery of the breast and axilar lymph node surgery with exercise of the upper limb and instruction to continue after discharge.
  Interventions: Other: PHYSICAL THERAPY
- Breast, axillar surgery without exercise (Active Comparator): The patients that underwent surgery of the breast and axilar nodes samples or dissection are discharged without exercise and instructions.
  Interventions: Other: PHYSICAL THERAPY

INTERVENTIONS:
Other: PHYSICAL THERAPY — EXERCISES AND EDUCATION TO FOLLOWING AFTER DISCHARGE PHYSICAL TREATMENT

SUMMARY:
Surgical treatments can cause late effects influencing activity of daily living, physical activity, and overall health. Late effects include persistent pain reported by 30 - 50% of women that underwent breast operations, restrictions of arm and shoulder movement were reported in 35% of patients, lymphedema in 15 - 25% of women who undergo axillary lymph node dissection and in about 6% of women who undergo sentinel lymph node biopsy. Lymphedema results in physical impairments including compromised function, diminished strength, fatigue, and pain in the affected arm . The axillary web syndrome is a self-limiting and frequently overlooked cause of significant morbidity in the early postoperative period after breast cancer, which is characterized by axillary pain that runs down the medial arm, limited shoulder range of motion (ROM) .

Physiotherapy and exercise in the postoperative period can result in a significant improvement in shoulder ROM in women treated for breast cancer, Additionally, exercises are an effective intervention to improve quality of life, cardiorespiratory fitness, physical functioning and fatigue in breast cancer patients. However, in the postoperative period consideration should be given to the early implementation of exercises because of the potential for seroma and increases in wound drainage volume and duration.

There is limited evidence on the influence of postoperative physiotherapy intervention, and instruction program on upper limb range of motion and return to physical activity divided by the type of surgery and regarding complications.

DETAILED DESCRIPTION:
Aim The aim of this study is to evaluate the influence of early postoperative physical therapy program on upper-limb function and returning to physical activity in the first 6 months following surgery.

Hypotheses

* Early physical activity performed post-operative will improve ROM and therefore, will help women after breast surgeries to return faster to their routine physical activity and by that promote physical health.
* Early postoperative physical therapy is safe when the program for is tailored to the type of surgery.

Methods

Study design Parallel group prospective randomized controlled clinical trial. Two surgical department's including general surgery department and genecology department in Assuta hospital, Tel Aviv, Israel

Sample All women undergoing breast cancer surgeries in Assuta hospital between 02.01.2018 and till 07.01.2019 will be randomized into two groups: Group A (intervention group) will be instructed first day post-operative to exercise program; Group B (control group) without intervention.

ELIGIBILITY:
Inclusion Criteria:

* Women
* Age 18-65.
* Diagnosed with breast cancer, undergoing breast surgery,
* Functional independence prior to the operation.
* Ability to communicate in Hebrew.

Exclusion Criteria:

* Cognitive disorders, patients unable to sign the consent form.
* Back and spinal morbidity.
* Fibromyalgia or chronic pain disorders.
* Neurological disorders.
* Renal failure with the need for dialysis.
* Lymphedema prior to surgery.
* History of breast surgery.
* Shoulder surgery or shoulder injuries with limited ROM.
* Ischemic heart disease, heart failure and radical heart insufficiency.
* Radical mastectomy, LD and DEIP reconstruction, exchange breast prosthesis.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female
Enrollment: 160 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2019-07-01 (Actual); Study Completion 2019-09-01 (Actual)

PRIMARY OUTCOMES:
Shoulder pain | 6 mnth
  The intensity of pain and chronological modification will be monitored

OTHER OUTCOMES:
Function of upper limb | six month
  The mobility of the shoulder will be evaluates in all movements
Complications | six month
  Possible complications after surgery will be recorded
Lymph edema | 6 mnth
  Radius of upper limb will be measured
physical activities influence in recovery after breast cancer surgery | 6 mnth
  patient will be agruped by intensity and frequency of PA

CONTACTS AND LOCATIONS:
Overall Officials: Sergio G Susmallian, MD, Study Director — Assuta Medical Center
Locations (1):
- Assuta Medican Center, Tel Aviv, Israel

IPD SHARING:
Plan to Share IPD: Yes
The patient will be evaluated after discharge by meetings or though video calls/
Supporting Information: Study Protocol, ICF, CSR
Time Frame: February 01 2019
Access Criteria: Physiotherapy after breast cancer surgery

REFERENCES:
- [Derived] Klein I, Kalichman L, Chen N, Susmallian S. A comprehensive approach to risk factors for upper arm morbidities following breast cancer treatment: a prospective study. BMC Cancer. 2021 Nov 20;21(1):1251. doi: 10.1186/s12885-021-08891-5. PMID 34800988